CLINICAL TRIAL: NCT03083119
Title: The Methylation Regulation Mechanism of Blood Stasis Relevant miRNA Expression on Coronary Heart Disease
Brief Title: Efficacy and Safety of Xuesaitong Soft Capsule for Coronary Heart Disease Unstable Angina
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jie Wang (Other)
Responsible Party: Sponsor-Investigator, Jie Wang, Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81473561
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Coronary Heart Disease; Unstable Angina
MeSH Terms: conditions — Coronary Disease; Angina, Unstable

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xuesaitong soft capsule group (Experimental): Patients who confirmed by coronary angiography and diagnosed blood stasis syndrome of coronary heart disease are given conventional Western medicine treatment and Xuesaitong soft capsule.
  Interventions: Drug: Xuesaitong soft capsule
- Placebo Comparator (Placebo Comparator): Patients who confirmed by coronary angiography and diagnosed blood stasis syndrome of coronary heart disease are given conventional Western medicine treatment and placebo.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Xuesaitong soft capsule — Panax Notoginseng Saponins, Specification:0.33 per bag, once take two pills and twice a day during a month.
  Arms: Xuesaitong soft capsule group
Drug: Placebo oral capsule — Xuesaitong soft capsule Placebo, soft capsule, once take two pills and twice a day during a month.
  Arms: Placebo Comparator

SUMMARY:
In this study, typical cases of coronary heart disease are selected. They will be intervened by Xuesaitong soft capsules to investigate efficacy and safety for Coronary Heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of coronary angiography unstable angina
* Clinical diagnosis of unstable angina
* Age of 30 to 75 years old
* Not use thrombolysis, dilate coronary drugs within two weeks
* Sign the consent

Exclusion Criteria:

* Severe valvular heart disease
* Insulin-dependent diabetes
* mental disease
* Combined with severe liver, kidney, hematopoietic system disorder
* Patients with malignant tumors
* Pregnancy or breast-feeding women
* Recent history of trauma
* Drug allergy

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2017-03-20 (Estimated); Primary Completion 2017-04-20 (Estimated); Study Completion 2017-08-20 (Estimated)

PRIMARY OUTCOMES:
major adverse cardiovascular events | 60 days
  death, myocardial infarction, hospitalization for unstable angina or stroke
Seattle Angina Questionnaire | 60 days
  to evaluate patients by Seattle Angina Questionnaire
blood stasis syndrome scale of Coronary heart disease angina pectoris | 60
  to evaluate patients by blood stasis syndrome scale of Coronary heart disease angina pectoris

SECONDARY OUTCOMES:
lipid | 60
  Triacylglyceride,total cholesterol, low densith lipoprotein, high densith lipoprotein

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, Principal Investigator — Guang Anmen Hospital
Locations (1):
- Guang Anmen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Duan L, Liu Y, Li J, Zhang Y, Dong Y, Liu C, Wang J. Panax notoginseng Saponins Alleviate Coronary Artery Disease Through Hypermethylation of the miR-194-MAPK Pathway. Front Pharmacol. 2022 Jun 16;13:829416. doi: 10.3389/fphar.2022.829416. eCollection 2022. PMID 35784716